CLINICAL TRIAL: NCT05072951
Title: An Adaptive Sample Collection to Evaluate a Biomarker for Kidney Transplant Rejection
Brief Title: Urine Biomarker for Kidney Transplant Rejection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Exosome Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECT2021-002
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Graft Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urine Biomarker for Kidney Transplant Rejection — Biomarker for active kidney transplant rejection.

SUMMARY:
An adaptive sample collection to support biomarker evaluation for kidney transplant rejection.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Kidney Transplant

Exclusion Criteria:

* Pediatric patients, under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and Female, at least 18 years of age with a kidney transplant prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Biospecimen collection | 3 years after last enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Kumar, Study Chair — Exosome Diagnostics, Inc.

IPD SHARING:
Plan to Share IPD: Undecided